CLINICAL TRIAL: NCT01436994
Title: A Randomised Study of Two Anti-thyroid Drug Treatment Regimens in Young People
Brief Title: Antithyroid Drug Treatment of Thyrotoxicosis in Young People
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Tim Cheetham, Dr Tim Cheetham, Newcastle-upon-Tyne Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NUTH 2759
Record Dates: First submitted 2011-08-18; First posted 2011-09-20 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Paediatric Thyrotoxicosis
Keywords: thyrotoxic; thyrotoxicosis; paediatric; endocrinology; block and replace; dose titration; carbimazole
MeSH Terms: conditions — Thyrotoxicosis; Bites and Stings | interventions — Dental Occlusion; Carbimazole; Propylthiouracil; Thyroxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Block and Replace (Active Comparator): Carbimazole is commenced in a dose of 0.75 mg/kg/day. The intention is to completely prevent endogenous thyroxine production. Thyroxine is then added in a replacement dose as the thyroid hormone levels fall into the lower half of the laboratory normal range. The principal measure of control during the first 6 months will be thyroid hormone levels rather than TSH.
  Interventions: Procedure: Block and Replace; Drug: carbimazole; Drug: propylthiouracil; Drug: thyroxine
- Dose Titration (Active Comparator): Carbimazole is commenced in a dose of 0.75 mg/kg/day until thyroid hormone levels fall into the local laboratory normal range. The dose is then reduced to 0.25 mg/kg/day with the intention of maintaining the euthyroid state. The principal measure of control during the first 6 months will be thyroid hormone levels rather than TSH.
  Carbimazole is the preferred treatment because of the increased risk of hepatotoxicity with propylthiouracil but patients who are treated with propylthiouracil can also be recruited and randomised. 1mg of carbimazole is approximately equivalent to 10 mg of propylthiouracil.
  Drug: Carbimazole 5mg and 20 mg tablets. Administered as a once or twice daily regimen with total daily dose adjusted according to prevailing biochemistry Drug: propylthiouracil 50 mg tablets administered once daily with the dose adjusted according to the prevailing biochemistry.
  Interventions: Procedure: Dose Titration; Drug: carbimazole; Drug: propylthiouracil

INTERVENTIONS:
Procedure: Block and Replace — The primary objective of treatment is to maintain a euthyroid state with TSH and thyroid hormone levels in the local laboratory normal range. Carbimazole is commenced in a dose of 0.75 mg/kg/day (propylthiouracil - for dose see below) with the aim being to completely preventing endogenous thyroxine production. Thyroxine is then added in a low replacement dose as the thyroid hormone levels fall into the lower half of the laboratory normal range. The principle measure of control during the first 6 months will be thyroid hormone levels rather than TSH. Carbimazole is the preferred treatment because of the increased risk of hepatotoxicity with propylthiouracil but patients who are treated with propylthiouracil can also be recruited and randomised. 1mg of carbimazole is approximately equivalent to 10 mg of propylthiouracil.
  Other Names: Carbimazole; propylthiouracil; thyroxine
  Arms: Block and Replace
Procedure: Dose Titration — The primary objective of treatment is to maintain a euthyroid state with TSH and thyroid hormone levels in the local laboratory normal range.
  Carbimazole is commenced in a dose of 0.75 mg/kg/day until thyroid hormone levels fall into the local laboratory normal range. The dose is then reduced to 0.25 mg/kg/day with the intention of maintaining a euthyroid state as reflected by a free thyroxine and TSH within the normal range.
  Most paediatricians in the UK commence thyrotoxic children on carbimazole rather than propylthiouracil. Carbimazole is the preferred treatment because of the increased risk of hepatotoxicity with propylthiouracil but patients who are treated with propylthiouracil can also be recruited and randomised. The guidelines detailed above can be used in the knowledge that 1mg of carbimazole is approximately equivalent to 10 mg of propylthiouracil.
  Other Names: carbimazole; propylthiouracil
  Arms: Dose Titration
Drug: carbimazole — Carbimazole 5mg and 20 mg tablets Administered as a once or twice daily regimen with total daily dose adjusted according to prevailing biochemistry
Drug: propylthiouracil — 50 mg tablets administered once daily with the dose adjusted according to the prevailing biochemistry
Drug: thyroxine — 25mcg, 50mcg and 100mcg tabletes administered once daily with the dose adjusted according to the prevailing biochemistry
  Arms: Block and Replace

SUMMARY:
The investigators aim to establish whether biochemical control during anti-thyroid drug therapy in young people with thyrotoxicosis varies depending upon whether a 'block and replace' or 'dose titration' regimen is used. The investigators will also assess remission rates and the frequency of side-effects in the two treatment groups.

DETAILED DESCRIPTION:
Thyrotoxicosis is an uncommon disorder in childhood and adolescence with a UK incidence around 1 per 100,000 (0-15 years). Most patients with thyrotoxicosis have Graves' disease which develops because of thyrotropin (TSH) receptor stimulation by autoantibodies. Patients with Hashimoto's thyroiditis can also be thyrotoxic in the early phase of the disease and occasionally thyrotoxicosis develops because of activating mutations of the TSH receptor. Many general paediatricians have experience of managing patients with thyrotoxicosis but national guidelines to assist in patient care have not been produced to date.

There is no ideal therapy for thyrotoxicosis in children and adolescents. The three treatment modalities for thyrotoxicosis - anti-thyroid drugs (ATD), surgery and radioiodine all have significant disadvantages. Particular considerations when managing young people include:

1. Low remission rates following a course of ATD.
2. Concerns about the morbidity associated with thyroidectomy.
3. Inadequate data regarding the long term safety of radioiodine.

Children and adolescents presenting with autoimmune thyrotoxicosis in the UK are usually treated with ATD from diagnosis for 1 - 4 years. Treatment is then stopped and patients who relapse return to ATD or are offered more definitive treatment with surgery or radioiodine. Life-long thyroid hormone replacement will be required if the thyroid gland is removed by surgery or ablated by radioiodine.

Excess thyroid hormone can have a major detrimental impact on cognitive function as well as cardiovascular and skeletal health. The maintenance of a clinically and biochemically euthyroid state is therefore highly desirable. There are two possible approaches when treating patients with ATD.

* 'Block and replace' (combined) therapy - where thyroid hormone production is prevented by ATD and thyroxine is then added in a replacement dose.
* 'Dose titration' (adaptive) therapy - where the dose of ATD is adjusted so that hormone production is normalised.

Both strategies are used by adult endocrinologists but it is unclear which of these approaches is the most appropriate in the young person.

Potential advantages of the 'block and replace' regimen include:

* Improved stability with fewer episodes of hyper or hypothyroidism.
* A reduced number of venepunctures and visits to hospital.
* Improved remission rates following a larger anti-thyroid drug dose.

Potential advantages of the dose titration approach include:

* Fewer side effects with a lower anti-thyroid drug dose
* Improved compliance on one rather than two medications. A meta-analysis conducted primarily in adult patients concluded that 'dose titration' was the most appropriate way to manage thyrotoxicosis because of fewer ATD-related side-effects although a group of authors subsequently highlighted significant limitations of this study.

This study is a prospective, multi-centre trial which aims to establish which regimen - block and replace or dose titration - is the most appropriate medical therapy for thyrotoxicosis during childhood and adolescence.

* Primary completion date changed from January 2019 to November 2014
* Study completion date changed from January 2019 to November 2015

ELIGIBILITY:
Inclusion Criteria:

1. All patients with thyrotoxicosis aged between 2 and 16 years at the time of diagnosis. Thyrotoxicosis will be diagnosed by the paediatrician on the basis of the clinical picture and the biochemistry (suppressed TSH with high thyroid hormone levels).
2. Child has consented/assented or consent via parent/guardian has been gained prior to any study specific procedures

Exclusion Criteria:

1. Known toxic adenoma / toxic hyperplasia (germline activating TSHR mutation).
2. McCune Albright Syndrome.
3. Previous episodes of Thyrotoxicosis..
4. Known allergic response to any of the study medication or ingredients as per SmPC.
5. Previous participation in this study.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2004-07; Primary Completion 2014-12 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Biochemical control as reflected by the stability of blood thyroid stimulating hormone (TSH) concentrations | 2.5 years
  For each patient, TSH will be determined at each visit: the primary outcome variable is obtained by measuring the proportion of TSH concentrations that are outwith the laboratory normal range (in calculating this value, determinations made within six months of diagnosis are ignored).

SECONDARY OUTCOMES:
Remission rates as defined by patients who are biochemically euthyroid at the end of the 4 year study period. | 4 years
  To establish whether the remission rates post therapy in young people with thyrotoxicosis are affected by treatment with a 'block and replace' or 'dose titration' regimen. This will be determined by determining the proportion of individuals who are in remission ie who are biochemically euthyroid off ATD-thyroid drug therapy at the end of the of the study period (4 years). The proportion of subjects in remission following block and replace therapy will therefore be compared with the proportion in remission following dose titration.
The frequency of adverse events on the 2 treatment regimens. | 3 years
  This will be reflected by the number of participants with adverse events and by the proportion of patients changing to a different treatment during the study period.
Additional measures of biochemical control. | 3 years
  A comparison of the mean and variability of TSH and thyroid hormone concentrations in the 2 treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Cheetham, Principal Investigator — Newcastle upon Tyne Hospiatls NHS Foundation Trust
Locations (18):
- United Kingdom (18):
  - Royal Aberdeen Children's Hospital, Aberdeen
  - Birmingham Children's Hospital, Birmingham
  - Addebrookes Hospital, Cambridge
  - Wales College of Medicine, Cardiff
  - University Hospital, Coventry
  - Ninewells Hospital, Dundee
  - Royal Hospital for Sick Children, Edinburgh
  - Royal Hospital for Sick Children, Glasgow
  - Hereford Hospital, Hereford
  - Crosshouse Hospital, Kilmarnock
  - Alder Hey Children's Hospital, Liverpool
  - St Bart's Hospital, London
  - St George's Hospital, London
  - Royal Manchester Children's Hospital, Manchester
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Norfolk & Norwich University Hospitals, Norwich
  - Oxford Radcliffe Hospitals, Oxford
  - Sheffield Children's Hospital, Sheffield

REFERENCES:
- See also: British Society for Paediatric Endocrinology and Diabetes supports this study — http://www.bsped.org.uk/